CLINICAL TRIAL: NCT05966246
Title: The Effect of Prucalopride Succinate on Gastrointestinal Motility After Laparoscopic Gastrectomy : Prospective Double Blind Case-control Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, In Gyu Kwon, Associate professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3-2021-0480
Record Dates: First submitted 2023-07-21; First posted 2023-07-28 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prucalopride succinate group (Experimental): Taking prucalopride succinate from the first day to the fifth day after surgery.
  Interventions: Drug: Arm I : Experimental (Prucalopride succinate group)
- Control (mosapride citrate) group (Placebo Comparator): Taking mosapride citrate from the first day to the fifth day after surgery.
  Interventions: Drug: Arm II : Control (Mosapride citrate group)

INTERVENTIONS:
Drug: Arm I : Experimental (Prucalopride succinate group) — Experimental group taking prucalopride succinate from day 1 to day 5 after surgery
  Arms: Prucalopride succinate group
Drug: Arm II : Control (Mosapride citrate group) — Control gourp taking mosapride citrate from day 1 day 5 after surgery
  Arms: Control (mosapride citrate) group

SUMMARY:
In order to improve postoperative ileus in patients undergoing gastrointestinal surgery, digestive medications and prokinetics have been routinely used. Among them, mosapride citrate is widely used as a representative drug, as it is a 5-hydroxytryptamine 4 receptor agonist that increases gastrointestinal motility.

Prucalopride succinate (dihydrobenzofurancarboxamide) is a type of 5-hydroxytryptamine 4 receptor agonist that has a higher affinity for the 5-HT4 receptor compared to mosapride (a benzamide derivative) which belongs to the same class of drugs. Prucalopride succinate has been demonstrated to increase both gastric and colonic motility through in vivo and in vitro studies. As mentioned earlier, it exhibits high specificity for the 5-HT4 receptor. The 5-HT4 receptor is not expressed in the gastric mucosa but is expressed at low concentrations in the small intestine, whereas it is highly expressed in the colonic mucosa. Therefore, prucalopride is widely used as a therapeutic agent for chronic constipation by increasing colonic motility. Furthermore, Prucalopride succinate stimulates the 5-HT4 receptors present in the nerve terminals of the myenteric plexus, promoting the release of acetylcholine. The released acetylcholine acts on α7nAch receptors located on the surface of enteric smooth muscle cells, inhibiting inflammatory responses and reducing postoperative ilues.

A randomized controlled trial (RCT) conducted on 110 patients who underwent gastrointestinal surgery demonstrated that prucalopride succinate showed significant improvement in gastrointestinal motility compared to the control group. Currently, mosapride citrate is widely used as a prokinetic agent in clinical practice. However, preliminary studies have shown no significant efficacy, and when comparing abdominal X-ray images taken on the third day after surgery, there is no significant difference compared to the placebo group. As a result, it can be observed that the recovery of gastrointestinal motility after surgery is not primarily due to small bowel motility but rather delayed gas passing caused by colon motility. Therefore, it can be assumed that using drugs that increase colon motility may be effective in improving gastrointestinal motility after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with gastric adenocarcinoma pathologically before surgery
2. Patients who underwent complete surgical resection (R0 resection)
3. Patients with an ASA score of 3 or less

Exclusion Criteria:

1. Patients over 80 years of age
2. Ascites or peritoneal metastasis
3. If you have intestinal obstruction before surgery
4. If chemotherapy was performed before surgery
5. If cancer other than gastric cancer is diagnosed
6. If there is a history of previous major intra-abdominal long-term surgery or abdominal radiation therapy
7. In case of liver failure or renal failure
8. Pregnant women
9. If it is judged that uncontrolled diabetes can affect intestinal function
10. If you have a stoma

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2022-01-25 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Quantitative intestinal motility measurement using radio-opaque markers | Every day from the 1st day to the 5th day after surgery

SECONDARY OUTCOMES:
Measurement of the amount of food intake, first flatus time and first defecation time | Every day from the 1st day to the 5th day after surgery
  1. Quantitatively compare and analyze the amount of food eaten in the test group and the control group.
  2. Compare the first flatus appearance time and first defecation time in the test group and the control group.

CONTACTS AND LOCATIONS:
Locations (1):
- GangnamSeverance Hospital, Seoul, South Korea